CLINICAL TRIAL: NCT03539068
Title: Online and Shared Decision-Making Interventions to Engage Service Men and Women in Post-Deployment Mental Health Care
Acronym: eSDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IIR 16-096
Record Dates: First submitted 2018-05-10; First posted 2018-05-29 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: PTSD; Depression; Substance Use Disorder; Traumatic Brain Injury
Keywords: Veteran; Mental Health; War; Shared decision-making; Access to care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Substance-Related Disorders; Brain Injuries, Traumatic; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: RCT- Screening, Shared-decision making intervention with Veteran and Providers using Agency for Healthcare Research and Quality (AHRQ) model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WEB-ED Only Control Arm (No Intervention): Veterans who screen positive on one or more mental health screens in WEB-ED will be eligible for RCT and those who consent and are randomly assigned to the no intervention control group will receive no further intervention but asked to participate in a subsequent study phase that addresses VA and post-deployment care access
- WEB-ED+ Treatment Arm (Experimental): Veterans who screen positive on one or more mental health screens in WEB-ED will be RCT-eligible. RCT-consenters randomly assigned to the WEB-ED+ Treatment are will receive:
  * eHealth interfaces tailored to Veterans' VA and MHV enrollment needs (links for electronic VA enrollment, MHV and MHV premium status enrollment).
  * Shared decision making (SDM) interfaces: Patient Decision aids (PTSD, depression, alcohol abuse); SDM educational video; videos).
  * Access to study staff available through a toll-free number to assist both Veterans and providers, including addressing questions, problem-solving about or assisting with stuck points (e.g. getting screening results to the provider).
  Interventions: Behavioral: WEB-ED+ Treatment Arm

INTERVENTIONS:
Behavioral: WEB-ED+ Treatment Arm — Veterans who screen positive on one or more mental health screens in WEB-ED will be RCT-eligible. RCT-consenters randomly assigned to the WEB-ED+ Treatment are will receive::
  * eHealth interfaces tailored to Veterans' VA and MHV enrollment needs (links for electronic VA enrollment, MHV and MHV premium status enrollment).
  * Shared decision making (SDM) interfaces: Patient Decision aids (PTSD, depression, alcohol abuse); SDM educational video; videos).
  * Access to study staff available through a toll-free number to assist both Veterans and providers, including addressing questions, problem-solving about or assisting with stuck points (e.g. getting screening results to the provider).
  Arms: WEB-ED+ Treatment Arm

SUMMARY:
OEF/OIF/OND war Veterans have unique post-deployment care needs that the VA is striving to understand and address. Unfortunately, there is a significant disparity in utilization of mental health (MH) care and VA access as most war Veterans don't seek needed care. New interventions are urgently needed to address disparities in post-deployment MH treatment engagement for war Veterans and to support VA's efforts to provide them with optimal access and care. Online health interventions have been shown to be preferred by OEF/OIF combat Veterans and have the potential to promote access to VA MH care. The investigators' research team has developed a web-based interface (WEB-ED) evolved by feedback from Veterans that screens for common post-deployment MH and readjustment concerns, provides tailored education about positive screens, and facilitates linkage to VA resources. Data from the investigators' prior studies demonstrate WEB-ED can be successfully implemented within VA and activate Veterans to seek needed care. Furthermore, emerging evidence indicates that when patients are educated about their health conditions and treatment alternatives using shared decision-making (SDM), increased treatment participation and adherence, and better health outcomes result. Next steps include: linking Veteran WEB-ED screening results to a VA secure network so that a provider can access the results; and integrating a SDM interface to promote Veteran-Provider partnerships in patient-centered care. This study will improve the investigators' understanding of the most effective methods to reduce barriers to enrollment in VA/MHV and transferring important medical information using My HealtheVet (MHV). Furthermore, it will provide important information regarding how WEB-ED results can enhance the capability of VA providers and transition patient advocates to use Veterans' screening results to triage and engage Veterans in patient-centered MH care and promote VA provider adoption of WEB-ED+ to facilitate patient engagement. Online screening, tailored education, and links to geographically accessible VA resources has been shown to be preferred by Veterans, providing recognition of treatable post-deployment MH concerns, and education that reduces stigma. This study builds upon and augments this prior work with research to understand and evaluate the processes needed to integrate WEB-ED+ into current VHA systems to support efficient care delivery, facilitate patient-centered care, and address unmet need for MH care while also resolving disparities in VA and VA MH care access and engagement for war Veterans. WEB-ED+'s use of shared decision making is a key component for promoting these benefits. WEB-ED+ represents a readily implementable and cost-effective intervention that, with partner collaboration, can be integrated into VA systems through MHV. Findings have important policy implications for several operational partners heavily invested in the improved access and delivery of evidence-based mental health care for war Veterans.

DETAILED DESCRIPTION:
OEF/OIF/OND war Veterans have unique post-deployment care needs that the VA is striving to understand and address. Unfortunately, there is a significant disparity in utilization of mental health (MH) care and VA access as most war Veterans don't seek needed care. New interventions are urgently needed to address disparities in post-deployment MH treatment engagement for war Veterans and to support VA's efforts to provide them with optimal access and care. Online health interventions have been shown to be preferred by OEF/OIF combat Veterans and have the potential to promote access to VA MH care. The investigators' research team has developed a web-based interface (WEB-ED) evolved by feedback from Veterans that screens for common post-deployment MH and readjustment concerns, provides tailored education about positive screens, and facilitates linkage to VA resources. Data from the investigators' prior studies demonstrate WEB-ED can be successfully implemented within VA and activate Veterans to seek needed care. Furthermore, emerging evidence indicates that when patients are educated about their health conditions and treatment alternatives using shared decision-making (SDM), increased treatment participation and adherence, and better health outcomes result. Next steps include: linking Veteran WEB-ED screening results to a VA secure network so that a provider can access the results; and integrating a SDM interface to promote Veteran-Provider partnerships in patient-centered care. The investigators propose a three phase study to address the investigators' aims. Aim 1 (phase 1) the investigators will gather qualitative information from key VA and Veteran informants to create an enhanced version (WEB-ED+) of the investigators' Current WEB-ED that includes an eHealth and SDM interface. Aim 2 (phase 2) will use a randomized controlled trial (RCT) to test WEB-ED+ vs. Current WEB-ED in promoting VA MH care engagement. Aim 3 (phase 3) the investigators will employ a process evaluation to determine the feasibility and acceptability of WEB-ED+ for both Veterans and VA practitioner and to document the VA processes Veterans use to enroll and engage in VA MH care. This study will improve the investigators' understanding of the most effective methods to reduce barriers to enrollment in VA/MHV and transferring important medical information using My HealtheVet (MHV). Furthermore, it will provide important information regarding how WEB-ED results can enhance the capability of VA providers and transition patient advocates to use Veterans' screening results to triage and engage Veterans in patient-centered MH care and promote VA provider adoption of WEB-ED+ to facilitate patient engagement. Online screening, tailored education, and links to geographically accessible VA resources has been shown to be preferred by Veterans, providing recognition of treatable post-deployment MH concerns, and education that reduces stigma. This study builds upon and augments this prior work with research to understand and evaluate the processes needed to integrate WEB-ED+ into current VHA systems to support efficient care delivery, facilitate patient-centered care, and address unmet need for MH care while also resolving disparities in VA and VA MH care access and engagement for war Veterans. WEB-ED+'s use of shared decision making is a key component for promoting these benefits. WEB-ED+ represents a readily implementable and cost-effective intervention that, with partner collaboration, can be integrated into VA systems through MHV. Findings have important policy implications for several operational partners heavily invested in the improved access and delivery of evidence-based mental health care for war Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veterans returning from deployment to Iraq or Afghanistan within the prior 5 years who are residing in identified study states.

Exclusion Criteria:

* Disabilities that would adversely impact ability to independently complete online screening or not allow to talk on telephone.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1312 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne G. Sadler, PhD RN, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1312 completed WEB-ED, 1234 had positive screens, 996 were excluded for a number of reasons, 316 were consented and randomized.
Period: Overall Study
Arm/Group | WEB-ED+ Treatment Arm | WEB-ED Only Control Arm
Started | 214 | 102
Completed | 199 | 102
Not Completed | 15 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WEB-ED+ Treatment Arm | WEB-ED Only Control Arm | Total
Number analyzed (Participants) | 214 | 102 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.99 (10.04) | 45.56 (11.33) | 44.49 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 56 | 157
  Male | 113 | 46 | 159
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Five participants did not report race/ethnicity.
  Participants
    Race/Ethnicity: number analyzed (Participants) | 211 | 100 | 311
    Race/Ethnicity: White | 143 | 66 | 209
    Race/Ethnicity: African American | 20 | 14 | 34
    Race/Ethnicity: Hispanic | 20 | 3 | 23
    Race/Ethnicity: Other | 7 | 6 | 13
    Race/Ethnicity: Multirace | 21 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: VA Mental Health Treatment Engagement Validated by Self Report or VA Electronic Medical Record Review.
Description: VA mental health care appointment(s) in any VA clinic with a VA mental health care provider embedded in primary care or within mental health clinics: Both new and follow up
Time Frame: Within 1 year of Treatment Intervention
Measure: Count of Participants; unit: Participants
Arm/Group | WEB-ED+ Treatment Arm | WEB-ED Only Control Arm
Number analyzed (Participants) | 199 | 102
Participants | 98 | 7
Statistical Analysis 1: Comparison: WEB-ED+ Treatment Arm; Test type: Superiority; p < 0.00001, Chi-squared

2. Secondary Outcome: Shared Decision Making Interface Between VA Clinician and Veteran Validated by VA Electronic Medical Record Review
Description: Shared decision-making template use (specific to this study) by clinician participants validated by VA electronic medical record review.
Time Frame: Within 1 year of Treatment Intervention
Measure: Count of Participants; unit: Participants
Arm/Group | WEB-ED+ Treatment Arm | WEB-ED Only Control Arm
Number analyzed (Participants) | 199 | 102
Participants | 89 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study entry until the end of study participation, at WEB-ED completion for baseline, at RCT inclusion, and at final interview (an average of 8 months)
Arm/Group | WEB-ED+ Treatment Arm | WEB-ED Only Control Arm
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/214 | 0/102
Other Adverse Events (participants affected / at risk) | 0/214 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03539068/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03539068/ICF_001.pdf